CLINICAL TRIAL: NCT00105105
Title: A Double-blind, Placebo-controlled Trial of the Safety and Efficacy of C-1073 (Mifepristone) as Adjunctive Therapy in Alzheimer's Disease
Brief Title: Mifepristone as Adjunctive Therapy in Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Collaborators: Institute for the Study of Aging (ISOA) (Other)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0069
Record Dates: First submitted 2005-03-04; First posted 2005-03-07 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2005-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimers; cognition; acetyl cholinesterase inhibitor; GR-II antagonist
MeSH Terms: conditions — Alzheimer Disease | interventions — Mifepristone

INTERVENTIONS:
Drug: Mifepristone

SUMMARY:
The purpose of this study is to evaluate the effects of C-1073 (Mifepristone) on cognition in patients with Alzheimer's disease (AD) who are also taking an acetylcholinesterase inhibitor (Aricept, Exelon or Reminyl).

DETAILED DESCRIPTION:
This will be a double blind, placebo controlled study of C-1073 to evaluate the effects on cognition in patients with mild to moderate Alzheimer's disease who are already receiving an acetylcholinesterase inhibitor and have been on a stable dose for at least 12 weeks. Patients will be randomized (1:1) to either daily dosing with 300 mg C-1073 or a placebo for 16 weeks. Patients will continue the stable daily dose of acetylcholinesterase inhibitor throughout the study.

Visits will be weekly at the beginning of the study, then every two weeks, and every 4 weeks after week 12. Assessments during these visits may include cognition and behavior, depression, safety, as well as physical exams, clinical laboratory tests, EKG and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease
* Women must have had a partial or complete hysterectomy
* Mini Mental Status Evaluation score of 18-27
* HAM-D score less than or equal to 18
* Able to provide written informed consent
* On a stable dose of an acetylcholinesterase inhibitor for at least 12 weeks prior to screening visit
* Ambulatory, or ambulatory with walker or cane
* Sufficient hearing and vision to enable the patient to comply with the study procedures
* Caregiver available to participate in the assessment of the patient and monitor dosing

Exclusion Criteria:

* Women with an intact uterus
* A clinically significant medical condition, including lab abnormality, which in the opinion of the investigator would place the patient at undue risk, or would impair the patient's ability to participate in the study. These include but are not limited to: history of cerebral vascular accident (CVA), adrenal insufficiency, porphyrias, autoimmune disorders, type I diabetes, chronic obstructive pulmonary disease (COPD), hematologic or oncologic disorders in the previous 2 years, vitamin B12 or folate deficiency
* A clinically significant active gastrointestinal, renal, hepatic, endocrine, or cardiovascular system disease that is not well controlled by diet, pharmacological treatment, or other therapeutic intervention
* History of psychotic episodes or bipolar disorder, or additional diagnosis of delusions, delerium, or depression
* Evidence of other psychiatric or neurologic disorders (e.g., stroke, schizophrenia, or Parkinson disease)
* Hachinski ischemia score of 5 or more
* Known hypersensitivity to cholinesterase inhibitors
* Use of systemic or pulmonary inhaled corticosteroids within the 30 days prior to randomization, or require use of these medications during the study
* Use of memantine (Namenda) within the 30 days prior to randomization, or require use of this medication during the study
* Currently taking medications known to significantly induce or inhibit the metabolism of CYP 3A4, or have taken these medications 7 days prior to randomization (see list below under prohibited medications)
* Use of anticholinergic compounds within the 30 days prior to randomization, or require use of this medication during the study
* History of electroconvulsive therapy (ECT); patients may not undergo ECT during the course of the trial
* Positive urine drug screen for any non-prescribed drug of abuse (including but not limited to amphetamines, cannabinoids, barbiturates, cocaine, opiates, benzodiazepines)
* History of illicit drugs usage or a history of drug or alcohol dependence
* Known to have another form of dementia that may also explain the patient's deficits including reversible dementias, Binswanger's, Parkinson's dementia complex, Korsakoff's, mental retardation or vascular dementia. Patients who meet clinical criteria for AD but who have deep white matter lesions on MRI or CT scan will be accepted.
* Currently taking prescription anticoagulants such as warfarin (Coumadin)
* Planned surgical procedures during the study period, including the 4 week off drug period between weeks 16 and 20
* Participation in a clinical investigation of any drug, or other biological or investigational therapy within 30 days prior to dosing
* Previous participation in a trial using mifepristone, or known sensitivity or allergy to C-1073 (mifepristone) or its constituents
* Body Mass Index (BMI) over 35

Prohibited Medications:

Medications known to significantly induce or inhibit the metabolism of CYP 3A4, specifically:

* carbamazepine (Carbatrol® Tegretol®)
* modafinil (Provigil®)
* nefazodone (Serzone®)
* droperidol
* erythromycin
* fluconazole (Diflucan®)
* itraconazole (Sporanox®)
* ketoconazole (Nizoral®)
* simvastatin (Zocor®)
* lovastatin (Mevacor®)
* vinblastine
* vincristine
* paclitaxel (Taxol®)
* tamoxifen (Nolvadex®)
* cyclosporine (Neoral®, Sandimmune®)
* tacrolimus (Gengraf®)
* sirolimus (Rapamune®)
* midazolam (Versed®)
* nicardipine (Cardene®)
* nifedipine (Adalat®, Procardia®)
* felodipine (Lexxel®, Plendil®)
* thioridizine
* pimozide (Orap®)
* quinidine
* Patient may also not take St. John's Wort during the study or within 7 days prior to study entry
* the use of grapefruit juice will be excluded during the course of the study.
* use of anticholinergic compounds over the past 30 days prior to randomization
* warfarin (Coumadin)
* all systemic and inhaled pulmonary corticosteroids
* memantine (Namenda)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 2003-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
effects on cognition

SECONDARY OUTCOMES:
effects on behavior and activities of daily living

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Pivotal Research Center, Mesa, Arizona
  - Pivotal Research Center, Peoria, Arizona
  - ATP Clinical Trials, Fountain Valley, California
  - UCI Irvine Medical Center, Orange, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - AVI Clinical Research, Torrance, California
  - Baumel-Eisner Neuromed Inst, Boca Raton, Florida
  - Baumel-Eisner Neuromed Inst, Fort Lauderdale, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Baumel-Eisner Neuromed Inst, Miami Beach, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Johnnie B. Byrd, Sr. Alzheimer's Center & Research Inst, Tampa, Florida
  - Memory Enhancement Center, Long Branch, New Jersey
  - Eastside Medical Research, New York, New York
  - Neuro Center of Ohio, Toledo, Ohio
  - Pahl Pharmaceutical Research, LLC, Oklahoma City, Oklahoma
  - Clinical Pharmaceutical Trials, Inc., Tulsa, Oklahoma
  - Clinical Trials Research Services, Pittsburgh, Pennsylvania
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - International Clinical Research Associates, Richmond, Virginia
  - International Clinical Research Associates, Virginia Beach, Virginia

REFERENCES:
- [Background] Belanoff JK, Jurik J, Schatzberg LD, DeBattista C, Schatzberg AF. Slowing the progression of cognitive decline in Alzheimer's disease using mifepristone. J Mol Neurosci. 2002 Aug-Oct;19(1-2):201-6. doi: 10.1007/s12031-002-0033-3. PMID 12212781
- See also: Corcept Therapeutics — http://www.corcept.com